CLINICAL TRIAL: NCT01767636
Title: A Phase II Efficacy Trial of Pazopanib in Non-clear Cell Metastatic Renal Cell Cancer (mRCC) PINCR
Brief Title: Pazopanib Hydrochloride in Treating Patients With Metastatic Kidney Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC1152; NCI-2012-02027 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MC1152 (Other: Mayo Clinic); 11-003340 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2013-01-10; First posted 2013-01-14 (Estimated); Results first posted 2020-04-08 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Carcinoma of the Collecting Ducts of Bellini; Chromophobe Renal Cell Carcinoma; Kidney Medullary Carcinoma; Kidney Oncocytoma; Metastatic Renal Cell Cancer; Papillary Renal Cell Carcinoma; Recurrent Renal Cell Carcinoma; Sarcomatoid Renal Cell Carcinoma; Stage IV Renal Cell Cancer
MeSH Terms: conditions — Carcinoma, Renal Cell; Oncocytoma, renal | interventions — pazopanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (pazopanib hydrochloride) (Experimental): Patients receive pazopanib hydrochloride PO QD on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Pazopanib Hydrochloride

INTERVENTIONS:
Drug: Pazopanib Hydrochloride — Given PO
  Other Names: GW786034B; Votrient

SUMMARY:
This phase II trial studies how well pazopanib hydrochloride works in treating patients with kidney cancer that has spread to other places in the body (metastatic). Pazopanib hydrochloride may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Pazopanib hydrochloride may also stop the growth of kidney cancer by blocking blood flow to the tumor.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the efficacy of pazopanib hydrochloride (pazopanib) in non clear cell metastatic renal cell cancer patients as assessed by the overall survival rate at 12 months.

SECONDARY OBJECTIVES:

I. To determine the rates of best tumor response at the end of the first two treatment cycles of pazopanib in non clear cell metastatic renal cell cancer patients.

II. To determine the benefit of pazopanib in increasing progression free survival time.

III. To describe toxicity profile of pazopanib in non clear cell metastatic renal cell cancer patients.

OUTLINE:

Patients receive pazopanib hydrochloride orally (PO) once daily (QD) on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Histological confirmation of non-clear cell renal cancer (including chromophilic [papillary], chromophobic, oncocytic, sarcomatoid, collecting duct [Bellini's duct]), translocation-type carcinoma or medullary renal cell carcinoma
* Up to one prior treatment for metastatic non clear cell carcinoma is allowed prior to registration as long as the agent used to treat was not pazopanib
* Measurable or non-measurable metastatic disease
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0, 1 or 2
* Absolute neutrophil count (ANC) >= 1500
* Platelets (PLT) >= 100,000
* Hemoglobin (HgB) > 9.0 g/dL; NOTE: subjects may not have had a transfusion within 7 days of registration
* Total bilirubin < 1.5 x upper limit of normal (ULN); NOTE: concomitant elevations in bilirubin above 1.0 x ULN is not permitted
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 2.5 x ULN; NOTE: concomitant elevations in ALT/AST above 1.0 x ULN is not permitted
* Urine protein to creatinine ratio (UPC) < 1; NOTE: if UPC >= 1, then a 24-hour urine protein must be assessed; subjects must have a 24-hour urine protein value < 1 g to be eligible
* Prothrombin time (PT) or international normalized ratio (INR) =< 1.2 x ULN; NOTE: subjects receiving anticoagulant therapy are eligible if their INR is stable and within the recommended range for the desired level of anticoagulation
* A female is eligible to enter and participate in this study if she is of:

  * Non-childbearing potential (i.e., physiologically incapable of becoming pregnant), including any female who has had:

    * A hysterectomy
    * A bilateral oophorectomy (ovariectomy)
    * A bilateral tubal ligation
    * Is post-menopausal
    * Subjects not using hormone replacement therapy (HRT) must have experienced total cessation of menses for >= 1 year and be greater than 45 years in age, OR, in questionable cases, have a follicle stimulating hormone (FSH) value > 40 mIU/mL and an estradiol value < 40 pg/mL (< 140 pmol/L)
    * Subjects using HRT must have experienced total cessation of menses for >= 1 year and be greater than 45 years of age OR have had documented evidence of menopause based on FSH and estradiol concentrations prior to initiation of HRT
  * Childbearing potential, including any female who has had a negative serum pregnancy test, =< 7 days prior to registration
  * Agrees to use adequate contraception; acceptable contraceptive methods, when used consistently and in accordance with both the product label and the instructions of the physician, are as follows:

    * Complete abstinence from sexual intercourse for 14 days before exposure to investigational product, through the dosing period, and for at least 21 days after the last dose of investigational product
    * Oral contraceptive, either combined or progesterone alone
    * Intrauterine device (IUD) or intrauterine system (IUS) with a documented failure rate of less than 1% per year
    * Male partner sterilization (vasectomy with documentation of azoospermia) prior to the female subject's entry into the study, and this male is the sole partner for that subject
    * Double barrier method: condom and an occlusive cap (diaphragm or cervical/vault caps) with a vaginal spermicidal agent (foam/gel/film/cream/suppository)
* Subjects must provide written informed consent prior to performance of study-specific procedures or assessments, and must be willing to comply with treatment and follow-up; procedures conducted as part of the subject's routine clinical management (e.g., blood count, imaging study) and obtained prior to signing of informed consent may be utilized for screening or baseline purposes provided these procedures are conducted as specified in the protocol
* Willing to return to Mayo Clinic enrolling institution for follow-up

Exclusion Criteria:

* Any of the following:

  * Nursing women
  * Pregnant women
  * Men or women of childbearing potential who are unwilling to employ adequate contraception
* Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens
* Immunocompromised patients (other than that related to the use of corticosteroids) including patients known to be human immunodeficiency virus (HIV) positive
* Prior history of receiving pazopanib treatments
* Uncontrolled intercurrent illness including, but not limited to:

  * Ongoing or active infection
  * Symptomatic anemia, uncontrolled hypertension (defined as systolic blood pressure [SBP] of >= 140 mmHg or diastolic blood pressure [DBP] of >= 90mmHg)
  * Symptomatic congestive heart failure as defined by the New York Heart Association (NYHA); does not exclude class III congestive heart failure (CHF)
  * Previously treated with therapies that are known to negatively impact cardiac function (e.g. prior treatment with anthracyclines)
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Evidence of active bleeding or bleeding diathesis
  * Psychiatric illness/social situations that would limit compliance with study requirements
  * Or any other serious uncontrolled medical disorders in the opinion of the investigator
* History of cerebrovascular accident including transient ischemic attack (TIA), myocardial infarction, pulmonary embolism or untreated deep venous thrombosis (DVT), coronary artery bypass graft surgery within 6 months prior to registration; Note: subjects with recent DVT who have been treated with therapeutic anti-coagulating agents for at least 6 weeks are eligible
* Receiving any other investigational agent which would be considered as a treatment for the primary neoplasm
* Other active malignancy =< 5 years prior to registration; EXCEPTIONS: non-melanotic skin cancer or carcinoma-in-situ of the cervix; NOTE: if there is a history or prior malignancy, they must not be receiving other specific treatment for their cancer
* History or clinical evidence of central nervous system (CNS) metastases or leptomeningeal carcinomatosis, except for individuals who have previously-treated CNS metastases, are asymptomatic, and have had no requirement for steroids or anti-seizure medication for 6 months prior to first dose of study drug; screening with CNS imaging studies (computed tomography [CT] or magnetic resonance imaging [MRI]) is required only if clinically indicated or if the subject has a history of CNS metastases
* Clinically significant gastrointestinal abnormalities that may increase the risk for gastrointestinal bleeding including, but not limited to:

  * Active peptic ulcer disease
  * Known intraluminal metastatic lesion/s with risk of bleeding
  * Inflammatory bowel disease (e.g. ulcerative colitis, Crohn's disease), or other gastrointestinal conditions with increased risk of perforation
  * History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess =< 28 days prior to registration
  * Clinically significant gastrointestinal abnormalities that may affect absorption of investigational product including, but not limited to:

    * Malabsorption syndrome
    * Major resection of the stomach or small bowel
* Corrected QT interval (QTc) > 480 msecs using Bazett's formula
* Receiving any medications or substances with risk of torsades de pointes; Note: medications or substances on the list "Drugs with Risk of Torsades de Pointes" are prohibited; medications or substances on the list "Drugs with Possible or Conditional Risk of Torsades de Pointes" may be used while on study with extreme caution and careful monitoring
* Known endobronchial lesions and/or lesions infiltrating major pulmonary vessels and/or hemoptysis in excess of 2.5 mL (or one half teaspoon) =< 8 weeks of registration
* Treatment with any of the following anti-cancer therapies: radiation therapy, surgery or tumor embolization, chemotherapy, immunotherapy, biologic therapy, investigational therapy or hormonal therapy =< 14 days prior to registration
* Prior autologous or allogeneic organ or tissue transplantation
* Elective or planned major surgery to be performed during the course of the trial
* Receiving any medications or substances that are strong or moderate inhibitors of cytochrome P450, family 3, subfamily A, polypeptide 4 (CYP3A4); use of the strong or moderate inhibitors are prohibited =< 7 days prior to registration
* Receiving any medications or substances that are inducers of CYP3A4; use of inducers are prohibited =< 7 days prior to registration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2013-05-16 (Actual); Primary Completion 2019-02-02 (Actual); Study Completion 2021-01-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian Costello, M.D., Principal Investigator — Mayo Clinic
Locations (3):
- United States (3):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Mayo Clinic, Rochester, Minnesota

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Pazopanib Hydrochloride): Patients receive 800 mg pazopanib hydrochloride PO QD on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Treatment (Pazopanib Hydrochloride)
Started | 38
Completed | 35
Not Completed | 3

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Pazopanib Hydrochloride)
Number analyzed (Participants) | 35
Age, Continuous [Median (Full Range); unit: years] | 63 [26 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 22
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 30
  More than one race | 0
  Unknown or Not Reported | 0
ECOG Performance Score at baseline [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group PS Scale: 0)Fully active, able to carry on all pre-disease performance without restriction; 1)Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work; 2)Ambulatory and capable of all selfcare but unable to carry out any work activities. Up and about more than 50% of waking hours; 3)Capable of only limited selfcare, confined to bed or chair more than 50% of waking hours; 4)Completely disabled. Cannot carry on any selfcare. Totally confined to bed or chair.
  Participants
    0 | 21
    1 | 12
    2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival Rate at 12 Months
Description: Overall survival rate at 12 months is defined as the percentage of participants who are alive at 12 months.
Time Frame: 12 months
Population: Evaluable participants are included in this analysis.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Pazopanib Hydrochloride)
Number analyzed (Participants) | 35
percentage of participants | 65.7 [50.5 to 78.9]

2. Secondary Outcome: Number of Participants Experiencing at Least One Toxicity
Description: Number of participants experiencing at least one toxicity defined as a grade 3 or higher adverse event deemed at least possible related to treatment.
Time Frame: Up to 2 years
Population: Evaluable participants are included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Pazopanib Hydrochloride)
Number analyzed (Participants) | 35
Participants | 17

3. Secondary Outcome: Progression-free Survival
Description: Kaplan-Meier curve will be used to estimate progression-free survival time. Progression is defined as At least one of the following must be true:a. At least one new malignant lesion, which also includes any lymph node that was normal at baseline (< 1.0 cm short axis) and increased to ≥ 1.0 cm short axis during follow-up. b. At least a 20% increase in PBSD (sum of the longest diameter for all target lesions plus the sum of the short axis of all the target lymph nodes at current evaluation) taking as reference the MSD. In addition, the PBSD must also demonstrate an absolute increase of at least 0.5 cm from the MSD.
Time Frame: From registration to the earliest date documentation of disease progression or death, assessed up to 2 years
Population: Evaluable participants are included in this analysis.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Treatment (Pazopanib Hydrochloride)
Number analyzed (Participants) | 35
months | 7.5 [5.0 to 11.0]

4. Secondary Outcome: Overall Survival
Description: Overall survival is defined as the time from study registration to death date.
Time Frame: Up to 2 years
Population: Evaluable participants are included in this analysis.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Treatment (Pazopanib Hydrochloride)
Number analyzed (Participants) | 35
months | 18.9 [13.0 to NA] — The 90% confidence interval upper limit was not reached (i.e. below the level of detection).

5. Secondary Outcome: Number of Participants With Best Response in the First 2 Cycles
Description: The number of participants with Best tumor response in the first 2 cycles. Partial Response (PR): At least a 30% decrease in PBSD (sum of the longest diameter for all target lesions plus the sum of the short axis of all the target lymph nodes at current evaluation) taking as reference the BSD. Progression is defined as At least one of the following must be true:a. At least one new malignant lesion, which also includes any lymph node that was normal at baseline (< 1.0 cm short axis) and increased to ≥ 1.0 cm short axis during follow-up. b. At least a 20% increase in PBSD (sum of the longest diameter for all target lesions plus the sum of the short axis of all the target lymph nodes at current evaluation) taking as reference the MSD. In addition, the PBSD must also demonstrate an absolute increase of at least 0.5 cm from the MSD.Stable Disease (SD): Neither sufficient shrinkage to qualify for PR, nor sufficient increase to qualify for PD taking as reference the MSD.
Time Frame: Up to 56 days
Population: Evaluable participants are included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Pazopanib Hydrochloride)
Number analyzed (Participants) | 35
Participants
  Partial Response (PR) | 4
  Stable Disease (SD) | 21
  Progression (PD) | 3
  Not Evaluated | 7

ADVERSE EVENTS:
Time Frame: Up to 2 years
Arm/Group | Treatment (Pazopanib Hydrochloride)
All-Cause Mortality (participants affected / at risk) | 19/35
Serious Adverse Events (participants affected / at risk) | 10/35
Other Adverse Events (participants affected / at risk) | 34/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Pazopanib Hydrochloride) (N=35)
Hypothyroidism (Endocrine disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 4 (4)
Colonic obstruction (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorders - Oth spec (Gastrointestinal disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Pazopanib Hydrochloride) (N=35)
Anemia (Blood and lymphatic system disorders) | 3 (5)
Hypothyroidism (Endocrine disorders) | 4 (7)
Blurred vision (Eye disorders) | 1 (1)
Dry eye (Eye disorders) | 1 (1)
Watering eyes (Eye disorders) | 1 (2)
Abdominal pain (Gastrointestinal disorders) | 6 (7)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 23 (95)
Esophageal pain (Gastrointestinal disorders) | 1 (3)
Flatulence (Gastrointestinal disorders) | 2 (4)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorders - Oth spec (Gastrointestinal disorders) | 1 (1)
Gastroparesis (Gastrointestinal disorders) | 1 (2)
Mucositis oral (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 9 (20)
Vomiting (Gastrointestinal disorders) | 6 (8)
Edema limbs (General disorders) | 1 (1)
Fatigue (General disorders) | 31 (190)
Gen disord and admin site conds-Oth spec (General disorders) | 1 (2)
Pain (General disorders) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 1 (1)
Alanine aminotransferase increased (Investigations) | 23 (69)
Alkaline phosphatase increased (Investigations) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 18 (44)
Blood bilirubin increased (Investigations) | 5 (11)
CD4 lymphocytes decreased (Investigations) | 2 (2)
Creatinine increased (Investigations) | 3 (7)
Ejection fraction decreased (Investigations) | 2 (2)
INR increased (Investigations) | 1 (3)
Lymphocyte count decreased (Investigations) | 5 (13)
Neutrophil count decreased (Investigations) | 4 (6)
Platelet count decreased (Investigations) | 3 (15)
Weight loss (Investigations) | 3 (15)
White blood cell decreased (Investigations) | 7 (11)
Anorexia (Metabolism and nutrition disorders) | 6 (20)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 2 (2)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (2)
Hypomagnesemia (Metabolism and nutrition disorders) | 5 (8)
Hyponatremia (Metabolism and nutrition disorders) | 10 (17)
Hypophosphatemia (Metabolism and nutrition disorders) | 5 (9)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (4)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (2)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 5 (26)
Headache (Nervous system disorders) | 2 (3)
Paresthesia (Nervous system disorders) | 1 (3)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 4 (21)
Proteinuria (Renal and urinary disorders) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 1 (1)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (12)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Palmar-plantar erythrodysesthesia syndrm (Skin and subcutaneous tissue disorders) | 1 (2)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 (3)
Skin and subcut tissue disord - Oth spec (Skin and subcutaneous tissue disorders) | 4 (15)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 2 (8)
Hypertension (Vascular disorders) | 28 (149)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-08-07): https://cdn.clinicaltrials.gov/large-docs/36/NCT01767636/Prot_SAP_000.pdf
  • Informed Consent Form (2018-08-01): https://cdn.clinicaltrials.gov/large-docs/36/NCT01767636/ICF_001.pdf